CLINICAL TRIAL: NCT02504554
Title: Treating Gastrointestinal Problems in Children With Autism Using Beneficial Bacteria Treatment (BBT)
Brief Title: Beneficial Bacteria Treatment for Autism
Acronym: BBT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Northern Arizona University (Other); University of Arizona (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001053
Record Dates: First submitted 2015-03-30; First posted 2015-07-22 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Problems; Autism Spectrum Disorders
Keywords: children
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Vancomycin; MoviPrep; Omeprazole; Microscopy, Electron, Scanning Transmission; Freezing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Group (Experimental): This group will receive all treatments orally. The treatments include a combination of Vancomycin, MoviPrep, Prilosec, and human fecal material; processed, frozen.
  Interventions: Drug: oral Vancomycin; Drug: MoviPrep; Drug: Prilosec; Biological: human fecal material; processed, frozen administered orally
- Rectal Group (Experimental): This group will receive some treatments rectally and some orally. The treatments include a combination of Vancomycin, MoviPrep, Prilosec, and human fecal material; processed, frozen.
  Interventions: Drug: oral Vancomycin; Drug: MoviPrep; Drug: Prilosec; Biological: human fecal material; processed, frozen; administered orally and rectally

INTERVENTIONS:
Drug: oral Vancomycin — an antibiotic
Drug: MoviPrep — a bowel cleanse
Drug: Prilosec — a stomach acid suppressan
Biological: human fecal material; processed, frozen administered orally — human fecal material; processed, frozen, administered orally
  Arms: Oral Group
Biological: human fecal material; processed, frozen; administered orally and rectally — human fecal material; processed, frozen; administered orally and rectally
  Arms: Rectal Group

SUMMARY:
This is an open-label clinical trial to investigate a combination therapy for treating gastrointestinal problems in children with autism spectrum disorders.

The combination therapy includes beneficial bacteria.

DETAILED DESCRIPTION:
This is an open-label clinical trial to evaluate the safety, tolerability, and feasibility of a combination therapy to treat gastrointestinal problems in children with autism spectrum disorders.

It involves a combination therapy including beneficial bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 7-17 years
2. Diagnosis of autism per Autism Diagnostic Interview-Revised (ADI-R)
3. Moderate or Severe GI problems ( on the GSRS, a single score of 4 (severe) on any item, or a score of 3 (moderate) on two items, or a score of 2 (mild) or more on any 4 items
4. No changes in medications, supplements, diet, therapies, or education in last 3 months, and no intention to change them during clinical trial
5. General good physical health aside from gastrointestinal problems
6. Cognitive Ability to Provide Informed Assent

Exclusion Criteria:

1. Antibiotics in last 6 months
2. Probiotics in last 3 months
3. Single-gene disorder (Fragile X, etc.)
4. Major brain malformation
5. Tube feeding
6. Severe gastrointestinal problems that require immediate treatment (life-threatening)
7. Ulcerative Colitis, Crohn's Disease, diagnosed Celiac Disease, Eosinophilic Gastroenteritis, or similar conditions
8. Severely underweight/malnourished
9. Recent or scheduled surgeries
10. Current participation in other clinical trials

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James B Adams, PhD, Principal Investigator — Arizona State University

REFERENCES:
- [Result] Kang DW, Adams JB, Vargason T, Santiago M, Hahn J, Krajmalnik-Brown R. Distinct Fecal and Plasma Metabolites in Children with Autism Spectrum Disorders and Their Modulation after Microbiota Transfer Therapy. mSphere. 2020 Oct 21;5(5):e00314-20. doi: 10.1128/mSphere.00314-20. PMID 33087514
- [Result] Kang DW, Adams JB, Coleman DM, Pollard EL, Maldonado J, McDonough-Means S, Caporaso JG, Krajmalnik-Brown R. Long-term benefit of Microbiota Transfer Therapy on autism symptoms and gut microbiota. Sci Rep. 2019 Apr 9;9(1):5821. doi: 10.1038/s41598-019-42183-0. PMID 30967657
- [Result] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Group | Rectal Group
Started | 12 (1 participant was switched from the oral group to the rectal group due to nausea/vomiting.) | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One of the participants in the oral group changed to the rectal group after nausea/vomiting with the initial oral dose. So, 13/5 changed to 12/6
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Group | Rectal Group | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 6 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal Symptom Responsiveness Scale (GSRS)
Description: The GSRS is a measure of gastrointestinal symptoms. It includes 15 questions, rated on a Likert scale of 1-7, from no symptoms to severe symptoms, respectively (i.e., higher is worse). We report an average score for all 15 questions, so the possible range for the average score is also 1-7.
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on all participants, regardless of how the initial dose of bacteria was administered (oral or rectal).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Combined Group: Combination of both groups
Arm/Group | Combined Group
Number analyzed (Participants) | 18
units on a scale
  Baseline | 2.74 (0.57)
  10 weeks | 1.31 (0.45)
Statistical Analysis 1: Comparison: Combined Group; Wilcoxon signed rank analysis of symptoms at 10 weeks (end of treatment) vs. baseline; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — no adjustment for multiple hypothesis testing since this was an exploratory study. the p-value listed is the actual result from analysis of the study data

2. Secondary Outcome: Parent Global Impressions-Revised (PGI-R)
Description: The PGI-R is a rating of change of 18 autism symptoms compared to baseline, with each symptom rated on a Likert scale from -3 (much worse) to zero (no change) to +3 (much better). We report the average change of the 18 symptoms, so the possible range is from -3 to +3.
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on all participants regardless of how the initial dose of bacteria was administered.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Group
Number analyzed (Participants) | 18
units on a scale | 1.4 (0.9)
Statistical Analysis 1: Comparison: Combined Group; Test type: Other — paired 2-sided t-test comparing baseline and 10 weeks (end of treatment); p < 0.001, t-test, 2 sided — no adjustment for multiple comparisons; paired t-test, 2 sided

3. Secondary Outcome: Blood Safety Markers (Assessment of Blood Chemistry Panel and Complete Blood Count)
Description: Number of participants who had a clinically significant change in their blood safety markers (comprehensive metabolic panel including kidney/liver function and complete blood count with differential)
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on 18 participants, regardless of how the initial dose of bacteria was administered.
Measure: Number; unit: participants
Arm/Group | Combined Group
Number analyzed (Participants) | 18
participants | 0

4. Secondary Outcome: Childhood Autism Rating Scale (CARS)
Description: The CARS is an assessment of 15 autism-related symptoms. Each item is scored on a scale of 1 (no symptoms) to 4 (severe symptoms), and the scores for each symptom are summed to obtain a total score. So, the possible scores range from 15 to 60, with a higher score indicating greater severity.
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on all participants, regardless of how the initial dose of bacteria was administered.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Group
Number analyzed (Participants) | 18
units on a scale
  Baseline | 39.7 (5.5)
  10 weeks | 34.1 (4.7)
Statistical Analysis 1: Comparison: Combined Group; Wilcoxon signed-rank test comparing the baseline score vs. the score at 10 weeks (end of treatment); Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — no adjustment for multiple comparisons The p-value listed is the result for the actual analysis of the data

5. Secondary Outcome: Social Responsiveness Scale (SRS)
Description: The SRS is an assessment of social skills based on 65 items, where each item is scored on a range of 0 (no symptoms) to 3 (severe symptoms). The total score is a sum of the individual scores, so the total possible range is from 0 to 195, with a higher score indicating greater severity of symptoms.
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on 18 participants, regardless of how the initial dose of bacteria was administered.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Group
Number analyzed (Participants) | 18
units on a scale
  Baseline | 116.2 (24.9)
  10 weeks | 97.8 (27.9)
Statistical Analysis 1: Comparison: Combined Group; Wilcoxon signed-rank test comparing scores at baseline vs. 10 weeks (end of treatment); Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney) — no adjustment for multiple comparisons the p-value listed is the actual result for the study results

6. Secondary Outcome: Short Sensory Profile
Description: The Short Sensory Profile is an assessment of sensory problems.
  However, the data on this scale was not collected due to administrative error.
Time Frame: baseline and 10 weeks
Population: Due to a logistical error, this data was not collected
Arm/Group | Oral Group | Rectal Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Vineland Adaptive Behavior Scale (VABS)
Description: The VABS is an assessment of adaptive behaviors, and we analyzed it to determine the developmental age of the participants, with possible scores ranging from 0 years to 21 years.
Time Frame: baseline and 18 weeks (8 weeks after treatment stopped)
Population: We report the data on all participants, regardless of how they received the initial dose of bacteria.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Combined Group
Number analyzed (Participants) | 18
years
  Baseline | 5.39 (2.48)
  18 weeks | 6.84 (2.81)
Statistical Analysis 1: Comparison: Combined Group; 2-sided t-test comparing the group at baseline vs. 18 weeks (8 weeks after end of treatment); Test type: Other; p < 0.001, t-test, 2 sided — no adjustment for multiple comparisons the p-value listed is the actual result for the analysis of the study data

8. Secondary Outcome: Daily Stool Record (DSR)
Description: The DSR is a record of the type of stool that a participant had each day, using the Bristol Stool Form which ranges from 1 (very hard) to 7 (liquid). We then analyzed the data as % days of abnormal stools over a 14 day period, where an abnormal stool is defined as an unusually hard stool (types 1-2), unusually soft stool (types 6-7), or no stool that day. So, the possible range of % days of abnormal stools is from 0% to 100%, with a higher score indicating a more severe problem.
Time Frame: Baseline and 10 weeks (end of treatment)
Population: We report the data on all participants, regardless of how the initial dose of bacteria was administered.
Measure: Mean (Standard Deviation); unit: percentage of days with abnormal stool
Arm/Group | Combined Group
Number analyzed (Participants) | 18
percentage of days with abnormal stool
  Baseline | 62 (22)
  10 weeks | 34 (24)
Statistical Analysis 1: Comparison: Combined Group; Wilcoxon signed rank test was used to compare scores at baseline vs. at 10 weeks (end of treatment); Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney) — no adjustment for multiple comparisons

ADVERSE EVENTS:
Time Frame: During the 10 weeks of treatment, and the 8 weeks of follow-up (18 weeks total).
Groups:
- All Groups: We report the data on 18 participants, regardless of how the initial dose of bacteria was administered. The reason is that all but one of the adverse events occurred during the vancomycin phase, which was common to both groups, and occurred before the randomization to receive the microbiota either orally or rectally. The only exception is one participant who had initial nausea/vomiting upon receiving the initial oral dose of microbiota, and they were switched from the oral group to the rectal group, which they tolerated without incident. There were no adverse effects from the microbiota.
Arm/Group | All Groups
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Groups (N=18)
rash (Skin and subcutaneous tissue disorders) | 1 (1) — One participant experienced a rash on their body after taking the vancomycin (flavored with natural orange). The vancomycin was stopped, the rash disappeared, and a non-flavored vancomycin was then administered without adverse effect
nausea/vomiting (Gastrointestinal disorders) | 1 (1) — 1 participant experienced nausea and vomiting with the first of the high-dose microbiota. She was switched to the rectal group, which was tolerated without adverse effect
hyperactivity and/or irritability (Nervous system disorders) | 12 (12) — Within 1-4 days after the start of the vancomycin, 12 children with ASD had a temporary hyperactivity (7 cases) or tantrums/aggression (5 cases). The symptoms lasted 1-3 days in most cases, but one participant had symptoms lasting for 3 weeks.

LIMITATIONS AND CAVEATS:
Small study, open-label design, but able to demonstrate safety and possible efficacy.

Dosage and duration not optimized, so adjustments in dosage and/or duration may improve results.

Therapy involved 4 medications; not clear if all needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No